CLINICAL TRIAL: NCT00458484
Title: Evaluation of a Radio-Surgical Approach for the Treatment of Kidney Tumors in Poor Surgical Candidates
Brief Title: Radiosurgery in Treating Patients With Kidney Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE12806; P30CA043703 (NIH); CASE12806 (Other: Case Comprehensive Cancer Center); NCI-2010-01064 (Other: NCI/CTRP)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Results first posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Kidney Cancer
Keywords: stage I renal cell cancer; stage II renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Series 1: Stereotactic radiosurgery (Experimental): Series I: Radiation will be delivered in 4 fractions. The initial dose level will be 6 Gy per fraction to a total dose of 24 Gy in 4 fractions. Doses will be escalated at 2 Gy per fraction increments to 12 Gy per fraction to a total dose of 48 Gy.
  Interventions: Radiation: stereotactic radiosurgery; Procedure: Renal Biopsy; Procedure: Serum Blood Markers
- Series 2: Stereotactic radiosurgery (Experimental): Series II: The initial dose level will be 48 Gy to the target volume (tumor) in 3 fractions of 16 Gy per fraction. If acute toxicity is acceptable, then the next four patients will be escalated to 54 Gy in 3 fractions of 18 Gy. Finally if a dose limit has not been reached, the last group of four patients will be treated to 60 Gy in 3 fractions of 20 Gy each.
  Interventions: Radiation: stereotactic radiosurgery; Procedure: Renal Biopsy; Procedure: Serum Blood Markers

INTERVENTIONS:
Radiation: stereotactic radiosurgery — Series I: Radiation will be delivered in 4 fractions.
  Series II: Radiation will be delivered in 3 fractions.
Procedure: Renal Biopsy — At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
Procedure: Serum Blood Markers — ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of blood will be collected within 2 hours prior to and following completion of fractionated radiation therapy to assess the levels of MIF (both MIF-1 and MIF-2) and VEGF.

SUMMARY:
RATIONALE: Radiosurgery can send x-rays directly to the tumor and cause less damage to normal tissue.

PURPOSE: This phase I/II trial studies the side effects and best dose of giving stereotactic radiosurgery and to see how well it works in treating patients with kidney tumors who are poor candidates for surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate and compare the clinical safety of utilizing four different schemes of radiosurgical ablative techniques for treating poor surgical candidates with renal tumors.

Secondary

* To evaluate and compare the clinical and radiographic efficacy of four different schemes of radiosurgical ablation of renal tumors in poor surgical candidates.

Serum Blood Marker Objective:

* To determine if serum markers collected before and after radiation may give a predictive indication of tumor response.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients undergo placement of 2-3 fiducial markers in or near the renal tumor. Patients then undergo 4 fractions of stereotactic radiosurgery in the absence of disease progression or unacceptable toxicity. Treatment may repeat at 6 months if tumor is still present.

After radio-surgery, follow-up will be done at 1 , 3 and 6 months and then every 6 months post radiosurgery for a total of 36 months.

PROJECTED ACCRUAL: A total of 32 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is considered a poor surgical candidate for removal of renal mass as determined by anesthesiology pre-operative assessment or the surgical team, medical team. (No major psychiatric illnesses.)
* Patient is able to give and sign study specific informed consent
* No prior radiation to the treatment field
* Negative serum or urine pregnancy test within 72 hours prior to registration for women of childbearing potential
* Patient has a radiologically and /or pathologically confirmed diagnosis of a renal tumor
* Karnofsky status of ≥ 60%
* Signed study-specific informed consent prior to study entry

Exclusion Criteria:

* Any patient not meeting the eligibility criteria.
* Any patient with active connective tissue disease such as lupus, dermatomyositis.
* Any patient with active Crohn's disease or active ulcerative colitis.
* Major psychiatric illness, which would prevent completion of treatment or interfere with follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-02-20 (Actual); Primary Completion 2017-03-12 (Actual); Study Completion 2019-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Machtay, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - UH-Chagrin Highlands, Orange, Ohio
  - UH-Westlake, Westlake, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited local hospital from 2/2007 to 5/2017.
Groups:
- Series 1/Dose Level 1: Stereotactic Radiosurgery: Dose Level I: Radiation will be delivered in 4 fractions:
  6 Gy x 4 fractions: Total of 24 Gy
  Renal Biopsy: At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
  Serum Blood Markers: ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of b
- Series 1/Dose Level 2: Stereotactic Radiosurgery: Dose Level 2: Radiation will be delivered in 4 fractions:
  8 Gy x 4 fractions: Total of 32 Gy
  Renal Biopsy: At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
  Serum Blood Markers: ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of b
- Series 1/Dose Level 3: Stereotactic Radiosurgery: Dose Level 3: Radiation will be delivered in 4 fractions:
  10 Gy x 4 fractions: Total of 40 Gy
  Renal Biopsy: At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
  Serum Blood Markers: ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of b
- Series 1/Dose Level 4: Stereotactic Radiosurgery: Dose Level 4: Radiation will be delivered in 4 fractions:
  12 Gy x 4 fractions: Total of 48 Gy
  Renal Biopsy: At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
  Serum Blood Markers: ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of b
- Series 2/Dose Level 1: Stereotactic Radiosurgery: Dose Level I: Radiation will be delivered in 3 fractions:
  16 Gy X 3 fractions: Total of 48 Gy
  Renal Biopsy: At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
  Serum Blood Markers: ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of b
- Series 2/Dose Level 2: Stereotactic Radiosurgery: Dose Level 2: Radiation will be delivered in 3 fractions:
  18 Gy x 3 fractions: Total of 54 Gy
  Renal Biopsy: At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
  Serum Blood Markers: ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of b
- Series 2/Dose Level 3: Stereotactic Radiosurgery: Dose Level 3: Radiation will be delivered in 3 fractions:
  20 Gy x 3 fractions: Total of 60 Gy
  Renal Biopsy: At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
  Serum Blood Markers: ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of b
Period: Overall Study
Arm/Group | Series 1/Dose Level 1: Stereotactic Radiosurgery | Series 1/Dose Level 2: Stereotactic Radiosurgery | Series 1/Dose Level 3: Stereotactic Radiosurgery | Series 1/Dose Level 4: Stereotactic Radiosurgery | Series 2/Dose Level 1: Stereotactic Radiosurgery | Series 2/Dose Level 2: Stereotactic Radiosurgery | Series 2/Dose Level 3: Stereotactic Radiosurgery
Started | 4 | 6 | 3 | 6 | 4 | 5 | 3
Completed | 4 | 6 | 3 | 6 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Not eligible b/c prior radiation history | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who went on treatment.
Groups:
- Series 1/Dose Level 1: Stereotactic Radiosurgery: Series I: Radiation will be delivered in 4 fractions: 6 Gy x 4 fractions total dose of 24 Gy.
  Renal Biopsy: At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
  Serum Blood Markers: ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of blood will be collected within 2 hours prior to and following completion of fractionated radiation therapy to assess the levels of MIF (both MIF-1 and MIF-2) and VEGF.
- Series 1/Dose Level 2: Stereotactic Radiosurgery: Series I: Radiation will be delivered in 4 fractions: 8 Gy x 4 fractions total dose of 32 Gy.
  Renal Biopsy: At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
  Serum Blood Markers: ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of blood will be collected within 2 hours prior to and following completion of fractionated radiation therapy to assess the levels of MIF (both MIF-1 and MIF-2) and VEGF.
- Series 1/Dose Level 3: Stereotactic Radiosurgery: Series I: Radiation will be delivered in 4 fractions: 10 Gy x 4 fractions total dose of 40 Gy.
  Renal Biopsy: At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
  Serum Blood Markers: ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of blood will be collected within 2 hours prior to and following completion of fractionated radiation therapy to assess the levels of MIF (both MIF-1 and MIF-2) and VEGF.
- Series 1/Dose Level 4: Stereotactic Radiosurgery: Series I: Radiation will be delivered in 4 fractions: 12 Gy x 4 fractions total dose of 48 Gy.
  Renal Biopsy: At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
  Serum Blood Markers: ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of blood will be collected within 2 hours prior to and following completion of fractionated radiation therapy to assess the levels of MIF (both MIF-1 and MIF-2) and VEGF.
- Series 2/Dose Level 1: Stereotactic Radiosurgery: Series II: Radiation will be delivered in 3 fractions: 16 Gy x 3 fractions total dose of 48 Gy.
  Renal Biopsy: At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
  Serum Blood Markers: ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of blood will be collected within 2 hours prior to and following completion of fractionated radiation therapy to assess the levels of MIF (both MIF-1 and MIF-2) and VEGF.
- Series 2/Dose Level 2: Stereotactic Radiosurgery: Series II: Radiation will be delivered in 3 fractions: 18 Gy x 3 fractions total dose of 54 Gy.
  Renal Biopsy: At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
  Serum Blood Markers: ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of blood will be collected within 2 hours prior to and following completion of fractionated radiation therapy to assess the levels of MIF (both MIF-1 and MIF-2) and VEGF.
- Series 2/Dose Level 3: Stereotactic Radiosurgery: Series II: Radiation will be delivered in 3 fractions: 20 Gy x 3 fractions total dose of 60 Gy.
  Renal Biopsy: At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
  Serum Blood Markers: ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of blood will be collected within 2 hours prior to and following completion of fractionated radiation therapy to assess the levels of MIF (both MIF-1 and MIF-2) and VEGF.
- Total: Total of all reporting groups
Arm/Group | Series 1/Dose Level 1: Stereotactic Radiosurgery | Series 1/Dose Level 2: Stereotactic Radiosurgery | Series 1/Dose Level 3: Stereotactic Radiosurgery | Series 1/Dose Level 4: Stereotactic Radiosurgery | Series 2/Dose Level 1: Stereotactic Radiosurgery | Series 2/Dose Level 2: Stereotactic Radiosurgery | Series 2/Dose Level 3: Stereotactic Radiosurgery | Total
Number analyzed (Participants) | 4 | 6 | 3 | 6 | 4 | 4 | 3 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 4
  >=65 years | 4 | 6 | 3 | 5 | 3 | 3 | 2 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 1 | 0 | 1 | 1 | 8
  Male | 3 | 3 | 2 | 5 | 4 | 3 | 2 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 6 | 3 | 5 | 4 | 4 | 3 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 4
  White | 3 | 6 | 2 | 5 | 4 | 3 | 3 | 26
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 3 | 6 | 4 | 4 | 3 | 30

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Radiosurgery
Description: Dose escalation stops if 2/4 (50%) or 3/8 (37.5%) of participants experience DLTs in a given dose level cohort. The maximum tolerated dose will be one dose level below which the DLTs were exceeded.
Time Frame: once every 4 weeks
Population: All participants who received treatment.
Measure: Number; unit: Gy
Arm/Group | Series 1: Stereotactic Radiosurgery | Series 2: Stereotactic Radiosurgery
Number analyzed (Participants) | 19 | 11
Gy | 48 | 60

2. Secondary Outcome: Overall Survival
Description: Radiographic efficacy as measured by overall (percent of participants still alive after study completion)
Time Frame: at 36 months from start of therapy
Population: All participants who received treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Series 1/Dose Level 1: Stereotactic Radiosurgery | Series 1/Dose Level 2: Stereotactic Radiosurgery | Series 1/Dose Level 3: Stereotactic Radiosurgery | Series 1/Dose Level 4: Stereotactic Radiosurgery | Series 2/Dose Level 1: Stereotactic Radiosurgery | Series 2/Dose Level 2: Stereotactic Radiosurgery | Series 2/Dose Level 3: Stereotactic Radiosurgery
Number analyzed (Participants) | 4 | 6 | 3 | 6 | 4 | 4 | 3
percentage of participants | 75 | 100 | 33 | 66 | 66 | 100 | 66

3. Secondary Outcome: Progression-free Survival
Description: Percent of participants still alive and without tumor progression at study completion
Time Frame: at 36 months from start of therapy
Population: All participants who received treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Series 1/Dose Level 1: Stereotactic Radiosurgery | Series 1/Dose Level 2: Stereotactic Radiosurgery | Series 1/Dose Level 3: Stereotactic Radiosurgery | Series 1/Dose Level 4: Stereotactic Radiosurgery | Series 2/Dose Level 1: Stereotactic Radiosurgery | Series 2/Dose Level 2: Stereotactic Radiosurgery | Series 2/Dose Level 3: Stereotactic Radiosurgery
Number analyzed (Participants) | 4 | 6 | 3 | 6 | 4 | 4 | 3
percentage of participants | 75 | 100 | 33 | 66 | 33 | 100 | 66

4. Secondary Outcome: Freedom From Local Progression
Description: Radiographic efficacy as measured as measured by freedom from local progression (percent of participants without local progression or local recurrence after study completion)
Time Frame: at 36 months from start of therapy
Population: All participants who received treatment.
Measure: Number; unit: percent
Arm/Group | Series 1/Dose Level 1: Stereotactic Radiosurgery | Series 1/Dose Level 2: Stereotactic Radiosurgery | Series 1/Dose Level 3: Stereotactic Radiosurgery | Series 1/Dose Level 4: Stereotactic Radiosurgery | Series 2/Dose Level 1: Stereotactic Radiosurgery | Series 2/Dose Level 2: Stereotactic Radiosurgery | Series 2/Dose Level 3: Stereotactic Radiosurgery
Number analyzed (Participants) | 4 | 6 | 3 | 6 | 4 | 4 | 3
percent | 100 | 100 | 100 | 100 | 100 | 100 | 66

5. Secondary Outcome: Freedom to Distant Recurrence
Description: Radiographic efficacy as measured by distant recurrance (percent of participants without distant failure after study completion)
Time Frame: at 36 months from start of therapy
Population: All participants who received treatment.
Measure: Number; unit: percent
Arm/Group | Series 1/Dose Level 1: Stereotactic Radiosurgery | Series 1/Dose Level 2: Stereotactic Radiosurgery | Series 1/Dose Level 3: Stereotactic Radiosurgery | Series 1/Dose Level 4: Stereotactic Radiosurgery | Series 2/Dose Level 1: Stereotactic Radiosurgery | Series 2/Dose Level 2: Stereotactic Radiosurgery | Series 2/Dose Level 3: Stereotactic Radiosurgery
Number analyzed (Participants) | 4 | 6 | 3 | 6 | 4 | 4 | 3
percent | 100 | 100 | 100 | 100 | 75 | 100 | 100

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a ten year time period from study activation to study completion. AEs were collected over a 3 year time period for each participant while on study.
Groups:
- Series 1/Dose Level 1: Stereotactic Radiosurgery: Dose Level I: Radiation will be delivered in 4 fractions:
  6 Gy x 4 fractions: Total of 24 Gy
  Renal Biopsy: At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
  Serum Blood Markers: ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of blood will be collected within 2 hours prior to and following completion of fractionated radiation therapy to assess the levels of MIF (both MIF-1 and MIF-2) and VEGF.
- Series 1/Dose Level 2: Stereotactic Radiosurgery: Dose Level 2: Radiation will be delivered in 4 fractions:
  8 Gy x 4 fractions: Total of 32 Gy
- Series 1/Dose Level 3: Stereotactic Radiosurgery: Dose Level 3: Radiation will be delivered in 4 fractions:
  10 Gy x 4 fractions: Total of 40 Gy
- Series 1/Dose Level 4: Stereotactic Radiosurgery: Dose Level 4: Radiation will be delivered in 4 fractions:
  12 Gy x 4 fractions: Total of 48 Gy
- Series 2/Dose Level 1: Stereotactic Radiosurgery: Dose Level I: Radiation will be delivered in 3 fractions: 16 Gy X 3 fractions: Total of 48 Gy
  Renal Biopsy: At 6 months,an optional percutaneous renal biopsy will be obtained of the targeted tumor, under ultrasound (US) or CT guidance.
  Serum Blood Markers: ELISA blood testing just prior to and immediately following each daily radiation therapy session. Approximately 5cc of blood will be collected within 2 hours prior to and following completion of fractionated radiation therapy to assess the levels of MIF (both MIF-1 and MIF-2) and VEGF.
- Series 2/Dose Level 2: Stereotactic Radiosurgery: Dose Level 2: Radiation will be delivered in 3 fractions: 18 Gy X 3 fractions: Total of 54 Gy
- Series 2/Dose Level 3: Stereotactic Radiosurgery: Dose Level 3: Radiation will be delivered in 3 fractions: 20 Gy X 3 fractions: Total of 6 Gy
Arm/Group | Series 1/Dose Level 1: Stereotactic Radiosurgery | Series 1/Dose Level 2: Stereotactic Radiosurgery | Series 1/Dose Level 3: Stereotactic Radiosurgery | Series 1/Dose Level 4: Stereotactic Radiosurgery | Series 2/Dose Level 1: Stereotactic Radiosurgery | Series 2/Dose Level 2: Stereotactic Radiosurgery | Series 2/Dose Level 3: Stereotactic Radiosurgery
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/6 | 1/3 | 2/6 | 1/4 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/6 | 1/3 | 3/6 | 3/4 | 1/4 | 1/3
Other Adverse Events (participants affected / at risk) | 0/4 | 1/6 | 0/3 | 1/6 | 1/4 | 3/4 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Series 1/Dose Level 1: Stereotactic Radiosurgery (N=4) | Series 1/Dose Level 2: Stereotactic Radiosurgery (N=6) | Series 1/Dose Level 3: Stereotactic Radiosurgery (N=3) | Series 1/Dose Level 4: Stereotactic Radiosurgery (N=6) | Series 2/Dose Level 1: Stereotactic Radiosurgery (N=4) | Series 2/Dose Level 2: Stereotactic Radiosurgery (N=4) | Series 2/Dose Level 3: Stereotactic Radiosurgery (N=3)
junctional rhythm (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Death not associated with CTCAE term - Death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Death not associated with CTCAE term - Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Necrosis, GI - Colon/cecum/appendix (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcer, GI - Duodenum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain - Cardiac/heart (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain - Chest wall (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain-Head injury, head pain due to a fall. (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal/Genitourinary Urosepsis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Series 1/Dose Level 1: Stereotactic Radiosurgery (N=4) | Series 1/Dose Level 2: Stereotactic Radiosurgery (N=6) | Series 1/Dose Level 3: Stereotactic Radiosurgery (N=3) | Series 1/Dose Level 4: Stereotactic Radiosurgery (N=6) | Series 2/Dose Level 1: Stereotactic Radiosurgery (N=4) | Series 2/Dose Level 2: Stereotactic Radiosurgery (N=4) | Series 2/Dose Level 3: Stereotactic Radiosurgery (N=3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rigors/chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight loss (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
SKIN OTHER: RT LEG ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIVERTICULITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-upper (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain - Bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain - Abdomen NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pain - Head/headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incontinence, urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intra-operative injury - NERVES: Peripheral sensory NOS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT00458484/Prot_SAP_000.pdf